CLINICAL TRIAL: NCT05192681
Title: Tislelizumab Combined With Docetaxel for Cross-line Treatment of First-line Resistant Advanced NSCLC，a Phase II Clinical Study
Brief Title: Tislelizumab as Cross-line Treatment for Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCOG003
Record Dates: First submitted 2022-01-05; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-10

CONDITIONS: Advanced Non-small-cell Lung Cancer
MeSH Terms: interventions — tislelizumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab arm (Experimental): Tislelizumab: 200 mg, intravenous infusion, administered on the 1st day of each cycle, every 3 weeks Docetaxel: 60-75mg/m2 administered on the 1st day of each cycle, every 3 weeks Treatment until the disease progresses or intolerable side effects appear.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab in combination with docetaxel until the development of PD, unacceptable toxicities, withdrawal of informed consent, end of study, lost to follow-up, or death, whichever occurs first.
  Other Names: Docetaxel

SUMMARY:
This study is a single-arm, prospective, open phase II clinical study, exploring the efficacy and safety for advanced non-small cell lung cancer after progression of first-line Tislelizumab combined with chemotherapy and continuing Tislelizumab in combination with docetaxel. The primary study endpoint of this study is measured by progression-free survival (PFS).

1. Tislelizumab: The recommended dose is 200 mg/dose administered every three weeks on the first day of each cycle.
2. Docetaxel: 60-75 mg/m2 every 3 weeks, administered on day 1 of each cycle.
3. Treatment cycle: Tislelizumab in combination with docetaxel until the development of PD, unacceptable toxicities, withdrawal of informed consent, end of study, lost to follow-up, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced non-small cell lung cancer diagnosed by histology or pathology, and has progressed after first-line treatment with tislelizumab combined with platinum-containing dual-drug chemotherapy
2. Patients who have progressed after first-line tislelizumab treatment for more than 3 months
3. No EGFR, ALK gene mutations (the genetic test is not required for patients with lung squamous cell carcinoma)
4. At least one measurable lesion (RECIST standard version 1.1)
5. The expected survival period is ≥3 months
6. The ECOG-PS score is 0-2 points

Exclusion Criteria:

1. The tumor histology or cytology is confirmed to be mixed adenosquamous carcinoma or combined with small cell lung cancer
2. Known or suspected active autoimmune diseases
3. A history of immunodeficiency or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and history of allogeneic bone marrow transplantation
4. Interstitial lung disease, drug-induced pneumonia, radiation pneumonia requiring steroid therapy or clinical symptoms, active pneumonia or severe lung dysfunction
5. Symptomatic brain metastases
6. Those who are known or suspected to be allergic to test drugs and their excipients
7. Women who are pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | five to six months
  the PFS of Tislelizumab combining with Docetaxel

SECONDARY OUTCOMES:
Overall survival | ten to eleven months
  the OS of Tislelizumab combining with Docetaxel

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian cancer hospital, Fuzhou, Fujian, China